CLINICAL TRIAL: NCT05205122
Title: Evaluation of Primary Congenital Glaucoma Management at Asyut University Hospital
Brief Title: Evaluation of Primary Congenital Glaucoma at Asyut University Hospital
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Omar Abdelkarem Hasan (Other)
Responsible Party: Sponsor-Investigator, Omar Abdelkarem Hasan, resident, Assiut University
Organization: Assiut University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Congenital glaucoma
Record Dates: First submitted 2022-01-11; First posted 2022-01-24 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Primary Congenital Glaucoma
MeSH Terms: conditions — Hydrophthalmos | interventions — Mitomycin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Infants with primary congenital glaucoma (Experimental)
  Interventions: Procedure: Combined trabeculotomy-trabeculectomy with mitomycin C

INTERVENTIONS:
Procedure: Combined trabeculotomy-trabeculectomy with mitomycin C — Combined trabeculotomy-trabeculectomy with mitomycin C Will be done in all cases

SUMMARY:
Evaluation of the management of primary congenital glaucoma regarding the results of surgical intervention at Asyut University Hospital

ELIGIBILITY:
Inclusion Criteria:

Typical symptoms of epiphora , photophobia and blepharospasm Corneal diameter > 13 mm Increased ocular tension > 25 mmHg UGA using schiotz tonometer

Exclusion Criteria:

Infants with history of previous surgery Secondary glaucoma Glaucoma associated with other congenital anomalies

Ages: 1 Day to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
IOP follow up | 1 year
  postoperative measurment of Intra ocular pressure by shoitz tonometer